CLINICAL TRIAL: NCT03017053
Title: The Optimal Neck Treatments Strategy of Early Oral Cancer Based on Adverse Pathological Factor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Chenping Zhang, Principal Investigator,Head of Oral and Maxillofacial- Head and Neck Oncology, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15411950300
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Oral Cancer
Keywords: Neck dissection; Survival; Early oral cancer; Early oral cavity squamous cancer with node negative neck
MeSH Terms: conditions — Mouth Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy (Experimental): Primary surgery & Radiotherapy
  Interventions: Radiation: Radiotherapy
- Elective neck dissection (Active Comparator): Primary surgery & Elective neck dissection
  Interventions: Procedure: Elective neck dissection

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy after primary surgery in the treatment of early oral cancer based on adverse pathological factor
  Arms: Radiotherapy
Procedure: Elective neck dissection — Elective neck dissection after primary surgery in the treatment of early oral cancer based on adverse pathological factor
  Arms: Elective neck dissection

SUMMARY:
Cervical nodal metastasis is the most certain prognostic factor in oral cancer. Appropriate management of the neck is therefore of paramount importance in the treatment of oral cancer. However, there is still some controversy on the treatment of early maxillofacial malignancies. Currently, investigators have no accurate uniform treatment standards, including the National Comprehensive Cancer Network (NCCN) recommended between surgery and radiotherapy options. Clinical evaluation indicated that lymph node-negative patients eventually 25%-35% had cervical node metastasis. Therefore, for the majority of patients with true node-negative, preventive cervical lymph node dissection is obviously over-treatment, and lower quality of life. Radiotherapy can avoid such surgery.

DETAILED DESCRIPTION:
Objective: To evaluate the effect of radiotherapy on the neck of early oral cancer with poor pathologic factors.

This is a randomized, prospective, open, multicenter study. Intervention: Patients receive primary tumor resection followed by radiotherapy.

Control: Patients receive primary tumor resection with selective neck dissection.

Primary:

2 years neck control rates

Secondary:

Disease-free survival (1, 2, 3, 5 years) Overall survival (3, 5 years) Quality of life

Endpoint definition:

1 year, 2 years, 3 years, 5 years disease-free survival is defined as: patients proportion from the date of surgery completion to 1 year, 2 years, 3 years, 5 years did not find clear evidence of recurrence or metastasis.

3 years, 5 years overall survival is defined as: the proportion of patients who survived from the beginning of the study to the third and fifth year in the total enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document
2. Age≥ 18 and≤ 75 years
3. Clinical/ Histological/ cytological/ Imaging examination proven Oral/Oropharynx Squamous-cell carcinoma (Tongue, buccal mucosa, mouth floor, hard palate, Molar area), the depth of invasion > 4mm in preoperative assessment
4. In line with clinical stage I / II stage (T1-2 N0 M0; AJCC 2010) and receiving surgical resection
5. KPS≥ 70
6. Normal bone marrow reserve function and normal liver, kidney function
7. Expected survival period≥ 6 months

Exclusion Criteria:

1. Inability to provide an informed consent
2. Evidence of oral distant metastasis or other malignancies
3. The patient has received prior surgery for primary tumor or lymph node ( except for biopsy )
4. Prior radiotherapy for primary tumor
5. The patient has previously received anti-tumor biological targeted therapy
6. The patient has received chemotherapy or immunotherapy for primary tumors
7. Prior malignancy within the previous 5 years (except for cured skin basal cell carcinoma or cervical carcinoma in situ)
8. With 3-4 grad Allergy to any drug in the treatment
9. Peripheral neuropathy> 1 grade
10. Any unstable systematic disease (including active infection, uncontrolled high blood pressure, unstable angina, onset of angina within the last 3 months, congestive heart failure, myocardial infarction within the previous 12 months, severe arrhythmia needing drug treatment, liver, kidney or metabolic disease)
11. HIV positive
12. Chronic diseases requiring immune agents or hormone therapy
13. Pregnant or lactating women
14. Drug/alcohol abuse, psychological or spiritual illness that may interfere compliance to the study
15. Patients with epilepsy requiring medications (such as steroids or antiepileptic drugs)
16. The patient has participated in other experimental therapy studies within 30 days
17. Researchers believe that the situation is unsuitable for participation in the group

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2016-07; Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Neck control rates | 2 years

SECONDARY OUTCOMES:
Disease-free survival | 1 year
Disease-free survival | 2 years
Disease-free survival | 3 years
Disease-free survival | 5 years
Overall survival | 3 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Chenping ZHANG, Ph.D, Principal Investigator — Shanghai Ninth People's Hospital Shanghai, China, 200011
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No